CLINICAL TRIAL: NCT01346631
Title: The Impact of a Paleolithic Diet on Sperm Parameters for Men Suffering From Male Infertility
Brief Title: The Paleolithic Diet and Male Factor Infertility
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We didn't start the study
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Dr. Amir Weiss/Senior Doctor, Clalit Health Services
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0130-10-EMC
Record Dates: First submitted 2011-05-01; First posted 2011-05-03 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male | interventions — Diet, Paleolithic

ARMS (1):
- paleolithic diet (Experimental): Subjects will adhere to a paleolithic diet for the duration of three months
  Interventions: Other: paleolithic diet

INTERVENTIONS:
Other: paleolithic diet — The diet consists of unlimited quantities of meat and fish, fruits and vegetables, eggs, nuts and water. Foods to be avoided include grains, wheat products, legumes, soy, potatoes and corn, rice, legumes, processed meats, soft drinks, dairy products and sugar. Allowed in moderation include coffee, alcohol,cooking oil, honey, salt, dried fruit.

SUMMARY:
Prospective studies concerning diet and male fertility are lacking. Observational studies suggest that a diet rich in fruits, vegetables and meats may be associated with higher sperm counts. The investigators wanted to see if a "paleolithic diet" consisting of meat, fish, fruits vegetables and nuts and lacking grains, legumes and dairy products can improve sperm counts.

ELIGIBILITY:
Inclusion Criteria:

* men with male infertility
* willingness to make dietary change for three months
* willingness to be blinded to sperm test results until the end of the experiment

Exclusion Criteria:

* High fever or abdominal or scrotal surgery during three months prior to intervention
* Change in diet, drinking or smoking habits in three months prior to intervention
* regular consumption of more than two servings of alcohol a day
* background ailment preventing dietary change

Min Age: 18 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Sperm Parameters | 3 months
  volume, concentration, motility, morphology

SECONDARY OUTCOMES:
Biomedical Indexes | 3 months
  Weight, blood pressure, CBC, liver enzymes, kidney function, lipid prophile, fasting glucose, HgbA1c, CRP, Testosterone, LH, FSH, Estradiol, TSH, Prolactin.

CONTACTS AND LOCATIONS:
Locations (1):
- HaEmek Medical Center, Afula, Israel